CLINICAL TRIAL: NCT04769297
Title: Micro-Dose, Macro-Impact: Leveraging Psychedelics in Frontline Healthcare Workers During the COVID-19 Pandemic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Limbic Medical (Other)
Collaborators: Enovex Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM-LDK-001
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Acute Stress Disorder
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Intervention Model Description: Retrospective, Open-label chart review
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sublingual Micro-Dose Ketamine (Experimental): Ketamine micro-dose 37.5mg compounded sublingual daily administration
  Interventions: Drug: Sublingual Micro-Dose Ketamine

INTERVENTIONS:
Drug: Sublingual Micro-Dose Ketamine — daily micro-dosing of frontline healthcare workers suffering from acute stress disorder due to the COVID-19 pandemic

SUMMARY:
A retrospective chart review of an open-label trial of low-dose ketamine administered to front-line Healthcare workers who were identified as experiencing acute stress disorder due to the COVID-19 Pandemic.

DETAILED DESCRIPTION:
An investigation of a novel, off-label use of an FDA approved drug (ketamine) in a low(micro) dose sublingual formulation of ketamine provided to front-line healthcare workers who were identified as suffering from acute stress disorder.

The study was conducted completely virtually via real-time telemedicine for physician visits and via asynchronous interaction for outcomes data collection.

Patients self-referred to the study via email outreach, and diagnosis was confirmed by medically validated screening assessments and study physician confirmation.

Once treatment was initiated, patients were seen via live telemedicine every 40 days while treatment response/outcomes data was collected weekly and monthly.

Patients were treated up to 120 days.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age
2. Demonstrate capacity to consent to the study
3. A Frontline Health Care Worker-defined as any EMS personnel (firefighter, EMT, flight nurse, etc.), or any hospital-based worker (particularly in the ED, ICU, or OR) such as an RN, MD/DO, or non-clinical support staff (EVS, etc.)
4. Experiencing acute stress disorder as determined by clinically validated screening tools -

Exclusion Criteria:

1. Currently on prescription medications for psychiatric issues
2. Currently pregnant or breastfeeding or actively trying to get pregnant
3. History of seizure disorder, liver disease, or psychosis/mania
4. Uncontrolled Hypertension
5. Physician discretion: any condition deemed inappropriate that will increase the risk -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Patient self-reported outcome measure | up to 120 days
  Perceived Stress Scale
Patient self-reported outcome measure | up to 120 days
  15-Dimensional Health-Related Quality of Life Questionnaire 15-Dimensional Health-Related Quality of Life Questionnaire
Patient self-reported outcome measure | up to 120 days
  PCL-5 (PTSD checklist for DSM-5)
Patient self-reported outcome measure | up to 120 days
  Physical Health- NIH PROMIS Global
Patient self-reported outcome measure | up to 120 days
  Mental Health- NIH PROMIS Global
Patient self-reported outcome measure | up to 120 days
  Health Perception and Social Roles
Patient self-reported outcome measure | up to 120 days
  Doctor's Note
Patient self-reported outcome measure | up to 120 days
  NIH PROMIS CAT- Depression
Patient self-reported outcome measure | up to 120 days
  NIH PROMIS CAT Neuro-QOL-Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Andre Atoian, MD, Principal Investigator — Limbic Medical
Locations (1):
- Limbic Medical, Toluca Lake, California, United States